CLINICAL TRIAL: NCT02267122
Title: Total Occlusive Ionic Silver-containing Dressing vs Mupirocin Ointment Application vs Conventional Dressing in Elective Colorectal Surgery: Effect on Incisional Surgical Site Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital General Universitario Elche (Other)
Responsible Party: Principal Investigator, Jaime Ruiz-Tovar, MD, PhD, Coordinator of Surgical Site Infections, Hospital General Universitario Elche
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Hospital General Elche
Record Dates: First submitted 2014-10-14; First posted 2014-10-17 (Estimated); Last update posted 2014-10-17 (Estimated); Status verified 2014-10

CONDITIONS: Incisional Surgical Site Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- ionic silver-containing dressing (Experimental): After placing the staples, a ionic silver-containing dressing was placed covering the wound.
  Interventions: Procedure: ionic silver-containing dressing
- Mupirocin ointment application (Experimental): After placing the staples, a Mupirocin ointment application was placed covering the wound.
  Interventions: Procedure: Mupirocin ointment application
- Conventional dressing (No Intervention): After placing the staples, a conventional dressing, without application of any special gauze or ointment, was placed covering the wound

INTERVENTIONS:
Procedure: ionic silver-containing dressing — After placing the staples, a ionic silver-containing dressing was placed covering the wound
  Arms: ionic silver-containing dressing
Procedure: Mupirocin ointment application — After placing the staples, Mupirocin ointment application over the wound was performed
  Arms: Mupirocin ointment application

SUMMARY:
The patients were randomized into 3 groups: those patients undergoing a ionic silver-containing dressing (ISD) (Group 1), those undergoing a Mupirocin ointment application (MOA) (Group 2) and those using a conventional dressing (Group 3) in the surgical wound after finishing an elective colorectal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of colorectal neoplasms and plans to undergo an elective surgery with curative aims.
* Open surgical approach

Exclusion Criteria:

* Anastomotic leak
* Mortality
* Lost to follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2012-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Incisional Surgical site infection | 30 postoperative days

REFERENCES:
- [Derived] Ruiz-Tovar J, Llavero C, Morales V, Gamallo C. Total Occlusive Ionic Silver-Containing Dressing vs Mupirocin Ointment Application vs Conventional Dressing in Elective Colorectal Surgery: Effect on Incisional Surgical Site Infection. J Am Coll Surg. 2015 Aug;221(2):424-9. doi: 10.1016/j.jamcollsurg.2015.04.019. Epub 2015 Apr 28. PMID 26206641